CLINICAL TRIAL: NCT05054608
Title: Long Term Outcome in ICU Treated COVID-19: Return to Work
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Dalarna County Council, Sweden (Other)
Responsible Party: Sponsor
Other Study IDs: U1111-1269-5745
Record Dates: First submitted 2021-09-20; First posted 2021-09-23 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Covid19
Keywords: Long term outcome; Return to work; COVID-19; Risk factors; Critical care
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 ICU cohort: All patients, 18 to 63 years old, admitted to a Swedish ICU with COVID-19 with at least one year of follow up. COVID-19 defined by the ICD-10 diagnosis U07.1 in the nationwide Swedish intensive care registry.
  Interventions: Other: No intervention
- COVID-19 hospital admission control cohort: Four random control patients per ICU patient matched on age legal gender and region. Controls selected from all patients admitted to a Swedish hospital with COVID-19 with at least one year of follow up. Not including patients in the COVID-19 ICU cohort. COVID-19 defined by the ICD-10 diagnosis U07.1 in the nationwide Swedish national patient registry.
  Interventions: Other: No intervention
- General population control cohort: Four general population controls per ICU patient, matched on age, legal gender and region drawn from the total population register of Sweden. Not including ICU and hospital admitted COVID-19 patients.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational study. No intervention.

SUMMARY:
Return to work (not being on sick leave) within one year after intensive care unit (ICU) admission with Coronavirus disease 2019 (COVID-19) will be assessed. Risk and risk factors for not having returned to work will be compared to patients admitted to hospital and general population controls.

The ICU population comprises all Swedish ICU patients with COVID-19 with at least one year of follow up. The hospital admitted cohort comprises four hospital admitted patients with COVID-19 per ICU patient, matched on age, legal gender and region. The general population controls are matched to the ICU patients in a one to four fashion on age, legal gender and region.

ICU patients are identified in the Swedish intensive care registry. The hospital admitted patients are identified in the national patient registry and the population controls are identified in the population registry. Data on socioeconomics and income are provided by the Statistics Sweden. Data on comorbidity, medications and death are provided from the National board of health and welfare. Finally, data on sick leave are provided from the Swedish Social Insurance Agency.

ELIGIBILITY:
Inclusion Criteria:

Admitted to a Swedish ICU and registered in the Swedish intensive care registry with the ICD 10 diagnosis U07.1 before 31 July 2020. ICU group.

or Admitted to hospital but not ICU with the ICD-10 diagnosis U07.1 in the national patient registry before 31 July 2020. Hospital group.

or randomly selected from the general population (and not included in the ICU or hospital admitted cohorts), matched on age, legal gender and region (four per ICU patient). Population control group

Exclusion Criteria:

Death within one year of inclusion. (For analysis of the secondary outcome). Missing a Swedish personal identification number

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of all patients a fulfilling the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 13537 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Is group an independent risk factor for having one or more additional sick leave free days alive? Ordinal logistic model including variables below. | One year
  Variables in binary logistic model: On sick leave one year before ICU admission, Charlson comorbidity index, age, legal gender, highest education, immigrant background, income the year before inclusion, marital status, group (ICU, Hospital or General population).

SECONDARY OUTCOMES:
Is cohort an independent risk factor for being on sick leave one year after inclusion? Binary logistic model containing the variables below? | One year
  Variables in linear regression model: On sick leave one year before ICU admission, Charlson comorbidity index, age, legal gender, highest education, immigrant background, income the year before inclusion, marital status, group (ICU, Hospital or General population).

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Lipcsey, Professor, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD sharing is not allowed under the ethical review approval.

REFERENCES:
- [Derived] Ahlstrom B, Frithiof R, Marks-Hultstrom M, Larsson IM, Strandberg G, Lipcsey M. The 1-Year Functional Recovery From Severe COVID-19 in a Swedish Working-Age Cohort. Acta Anaesthesiol Scand. 2025 Jul;69(6):e70058. doi: 10.1111/aas.70058. PMID 40356220